CLINICAL TRIAL: NCT00152308
Title: A Prospective, Placebo-Controlled, Double-Blind, Randomized Study Evaluating the Efficacy of Non-Polymer-Based Coating With Two Different Rapamycin-Dosages for the Prevention of Restenosis After Percutaneous Coronary Interventions
Brief Title: Non-Polymer-Based, Rapamycin-Eluting Stents to Prevent Restenosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrolement
Sponsor: Translumina GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GE IDE No. S01903
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2005-09

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Device: 2% rapamycin-eluting YUKONdes PEARL-stent
Device: 1% rapamycin-eluting YUKONdes PEARL-stent
Device: YUKONdes PEARL-stent coated with placebo (ethanol)

SUMMARY:
The purpose of the study is to evaluate the effectively of coating of coronary stents with two different doses of rapamycin for the prevention of coronary vessel re-blockage

DETAILED DESCRIPTION:
In-stent restenosis remains the major problem limiting the efficacy of coronary stenting. Either sirolimus or paclitaxel drug-eluting stents have been demonstrated to decrease neointima proliferation resulting in a remarkable reduction of restenosis rate. However, despite the outstanding results achieved with this novel approach to restenosis, some caveats still remain. Although sirolimus markedly decreased the restenosis rate among diabetic patients in SIRIUS trial, the benefit of treatment was modest in those diabetics treated with insulin as well as with lesions longer than 15 mm located in vessels smaller than 2.5 mm. Additionally, in a recent study it was reported that the restenosis rate in high-risk lesions such as coronary bifurcations still remains a problem Data from patient populations other than those enrolled in randomized trials suggest even more caution in the evaluation of the impact of DES on restenosis in the "real world", where the operator must deal with in-stent restenosis, bifurcation lesions, chronic total occlusions, small vessels, and long lesions. The identification of some of the traditional risk factors for restenosis as important predictors for in-DES restenosis could be explained as an insufficient inhibition of tissue reaction and neointimal growth by the antiproliferative action of the specific drug or dose used. This leads to the inference that an individualized approach should be adopted by tailoring the choice and the dosing of eluting drug(s) according to the specific lesion or patient characteristics. On the other hand, although drug-eluting stents are currently considered as the most effective way to reduce in-stent restenosis, their widespread use is hampered by the high costs. Therefore, it is important to develop new methods and techniques that would result in a more effective prevention of in-stent restenosis while being available for a larger number of patients. These considerations as well as the proven efficacy of rapamycin in lowering the rate of coronary restenosis, support the rationality of the concept of on-site coating of stents in the catheterization laboratory with individualized doses of rapamycin after the clinical and the angiographic profiles of the patient scheduled to coronary stenting have been determined

ELIGIBILITY:
Inclusion Criteria:

Age 18-85 years; Symptoms (stable or unstable angina) or signs of myocardial ischemia; Single de novo diagnosed lesion in a native coronary artery (50-99% DS); Lesion length 8 - 25 mm; Vessel diameter 2.25-3.75 mm; Written informed consent

Exclusion Criteria:

Left main target lesion unprotected by a graft; Ostial and bifurcation target lesion; Severely calcified lesions; Thrombus in target lesion; Tortuosity or angulation of target vessel or lesion; Treatment of nontarget lesions in the same or a different coronary vessel during the index procedure; Contraindications to the study medications; Acute myocardial infarction (< 48 h); Left ventricular ejection fraction < 25%; Participation in another trial; Pregnancy or lack of protection against pregnancy during the study Coexisting conditions limiting the life expectancy to less 24 months or that could affect the compliance of patients with protocol; Serum creatinin >2.0mg/dL; Hemorrhagic diathesis; Leukocyte count <3500/ml^3 Platelet count <100.000/ml^3

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2004-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Binary angiographic restenosis at follow-up angiogram

SECONDARY OUTCOMES:
Target vessel failure (all-cause death, myocardial infarction, or revascularization of the target lesion)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Kurt Huber, MD, Study Director — Wilhelminenspital der Stadt Wien
Locations (10):
- Austria (4):
  - St. Johanns Spital, Salzburg
  - Donauspital der Stadt Wien, Vienna
  - Allgemeines Krankenhaus Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- Germany (3):
  - Deutsches Herzzentrum Muenchen, Munich
  - Kardiologische Praxis und Praxisklinik, Munich
  - First Medizinische Klinik rechts der Isar, Munich
- Israel (3):
  - Hadassah University Hospital, Jerusalem
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Zrifin

REFERENCES:
- [Background] Hausleiter J, Kastrati A, Wessely R, Dibra A, Mehilli J, Schratzenstaller T, Graf I, Renke-Gluszko M, Behnisch B, Dirschinger J, Wintermantel E, Schomig A; investigators of the individualizable durg-eluting Stent System to Abrogate Restenosis Project. Prevention of restenosis by a novel drug-eluting stent system with a dose-adjustable, polymer-free, on-site stent coating. Eur Heart J. 2005 Aug;26(15):1475-81. doi: 10.1093/eurheartj/ehi405. Epub 2005 Jun 23. PMID 15975990
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Tanabe K, Serruys PW, Grube E, Smits PC, Selbach G, van der Giessen WJ, Staberock M, de Feyter P, Muller R, Regar E, Degertekin M, Ligthart JM, Disco C, Backx B, Russell ME. TAXUS III Trial: in-stent restenosis treated with stent-based delivery of paclitaxel incorporated in a slow-release polymer formulation. Circulation. 2003 Feb 4;107(4):559-64. doi: 10.1161/01.cir.0000048184.96491.8a. PMID 12566366